CLINICAL TRIAL: NCT01951404
Title: Does ALlopurinol Regress lefT Ventricular Hypertrophy in End Stage REnal Disease: The ALTERED Study
Acronym: Altered
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Dundee (Other)
Collaborators: British Heart Foundation (Other); NHS Tayside (Other Government); NHS Greater Glasgow and Clyde (Other); University of Glasgow (Other)
Responsible Party: Principal Investigator, Elaine Rutherford, Clinical Research Fellow - Principal Investigator, University of Dundee
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2012CV07
Record Dates: First submitted 2013-09-18; First posted 2013-09-26 (Estimated); Last update posted 2016-11-04 (Estimated); Status verified 2016-11

CONDITIONS: End Stage Renal Disease; Left Ventricular Hypertrophy
Keywords: Left Ventricular Hypertrophy; Allopurinol; End Stage Renal Disease; Haemodialysis; Renal Replacement Therapy; MRI
MeSH Terms: conditions — Kidney Failure, Chronic; Hypertrophy, Left Ventricular | interventions — Allopurinol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Allopurinol (Active Comparator): Participants in this arm will be given allopurinol with the dose gradually increasing weekly as tolerated up to the dose determined in the first phase of the study. The drug dose will be given orally 3 times weekly after dialysis for 1 year.
  Interventions: Drug: Allopurinol
- Placebo (Placebo Comparator): Participants in this arm will be given placebo with the dose appearing to gradually increase weekly as tolerated up to the dose determined in the first phase of the study. The drug dose will be given orally 3 times weekly after dialysis for 1 year.
  Interventions: Drug: Placebo (for allopurinol)

INTERVENTIONS:
Drug: Allopurinol
  Arms: Allopurinol
Drug: Placebo (for allopurinol)
  Arms: Placebo

SUMMARY:
Kidney patients on dialysis commonly die because of heart disease. One of the biggest problems in their hearts is that the muscle wall of the heart thickens. This makes it less efficient. We found in patients with mild kidney disease that a drug normally used to treat gout (allopurinol) had the remarkable side effect of being able to reduce this thickening of their heart wall. In this new study we aim to find out if this benefit of allopurinol also occurs in severe kidney patients i.e. those on regular dialysis. We also are trying to figure out the best dose of allopurinol to use. To do this we are planning a study where we will recruit patients with kidney disease who are on dialysis. The 1st phase of the trial will be to determine the best dose of allopurinol to use and the second phase will be to do a clinical trial where patients will be randomly allocated to either this optimum dose of allopurinol or a dummy medication (placebo) and will receive one year of treatment. They will have a special scan of the heart using an MRI machine to measure the extent of thickening of their heart muscle before they start on treatment and will have a further MRI scan when their one year treatment finishes.

Phase 1- the dose finding study, will involve 10 patients who will have between 3 and 7 visits to the hospital scheduled around 4 to 17 dialysis sessions. The later study will involve up to 76 patients who will be asked to attend the hospital up to 8 times over a 13 month period.

DETAILED DESCRIPTION:
The ALTERED trial is a randomised, double blinded, placebo controlled multi-centre study conducted in NHS Tayside, NHS Ayrshire & Arran & NHS Greater Glasgow & Clyde to compare allopurinol (dose to be confirmed from dose escalation study noted above) at either, 100mg, 200mg, 250mg, 300mg or 350mg to placebo.

Patients will be enrolled in this trial for a period of between 12 to 13 months.

At screening visit an initial history and clinical examination will be performed. Participants will then undergo an echocardiogram to ensure no significant heart failure unless they have had an ECHO in the previous 4 years..Should the participant be eligible for the study they will have a Cardiac Magnetic Resonance Imaging (MRI) scan prior to their baseline (Randomisation) visit. They will also have bloods taken for safety analysis, have a 12 lead ECG done, vital signs recorded and if they agree have 24 hour BP monitoring.

Once the patient is known to be eligible they will return - for the first randomisation, dosing visit at any time up to four weeks after screening. At this randomisation visit post dialysis session, eligible participants will be randomly assigned to either placebo or allopurinol 100mg.

They will continue on allopurinol/placebo 100mg for 2 weeks, with dosing after each dialysis session only. They can have FMD, PWV and PWA measurements taken. All participants will be offered the opportunity to opt in or out of the FMD, PWV and PWA measurements, which are secondary outcome measures only.

If study drugs are tolerated, the dose would be increased at weekly intervals after the 200mg dose to the allopurinol dose chosen by the dose escalation study, if greater than 200mg. Baseline blood samples will be taken for routine bloods including full blood count, renal function, liver function, random blood glucose, haemoglobin A1C, lipids, calcium and phosphate. These blood tests will be repeated at 6, 9 and 12 months. Routine safety bloods (including U+Es and LFTs) will be taken pre-dialysis at visits throughout the study. Subjects will be followed at baseline, week 2, week 6, month 6, month 9 and month 12. Research bloods and urate levels will be taken at baseline, week 6, months 6, 9 and 12. However, to ensure blinding throughout urate results will not be made available to the investigators until the end of the trial. BP is recorded as part of standard care and will be available for analysis. Pre and post-dialysis readings will be recorded. Other variables such as weight and fluid removed during dialysis are also noted as part of routine care and will be available for analysis. 24-hour BP will be performed at the start and end of the study if participants agree. Cardiac MRI scans will be performed at the start and at the end of the 12 month study period. Patients will continue with all their usual medication, which will remain unchanged throughout unless clinically indicated.

CMRI Methods The MRIs will normally be done on a non dialysis day. If this is not possible then we will rarely perform an MRI on a dialysis day. Baseline and repeat CMR examinations in screening (between 0-6 weeks before randomisation) and after the final 12 month (+/- 6 weeks) visit will be performed on similar 3T Magnetom scanners (Siemens, Erlangen, Germany) using dedicated phase array cardiac and phosphorous spectroscopy coils. Serial contiguous short-axis cines will be acquired from the vertical long axis and horizontal long axis of the left ventricle (electrocardiogram gated, steady-state free precession imaging [true fast imaging with steady-state precession], with the short axis imaging parameters being a repetition time of 2.5ms, echo time of 1.1ms, flip angle of 60°, and slice thickness 6mm). Analysis will be performed offline (Argus Software, Siemens) by a single blinded observer for the assessment of ventricular volumes (EDV, ESV, stroke volume), EF, and left ventricular mass. This single observer will analyse scans from both sites. The reproducibility of the left ventricular mass assessment using MRI will be derived for this observer. A test-retest intraobserver coefficient of variation of 2.0% is usual in our past MRI studies. We will also assess reproducibility between each site, although the same observer will assess all scans at both sites. We will take the opportunity to measure other MRI parameters of interest which are easily obtained with little extra scan time: Phosphorous -31 MR spectroscopy, T1 mapping and aortic compliance by methods already published by us.[29, 30] Both will give significant added value.

MR spectroscopy will see whether allopurinol increases high energy phosphates in ESRD (measured by PCr:ATP) which it is likely to do since it is known to increase ATP levels in vitro and it is now known to improve cardiac energetics (MRI measured) in human heart failure.[31, 32] We will measure high energy phosphates (HEP), comparing Phosphocreatine : Beta adenosine triphosphate (PCr:ATP) ratio from the long axis views of the left ventricle.[29] In addition we will use MRI to assess aortic vascular compliance and pulse wave velocity [30] using cine transverse thoracic aortic gated steady state free precession acquisitions which will complement well the other peripheral vascular measures of endothelial/vascular function being assessed (see below). Should a scanner at any site become unavailable for a prolonged period of time during the study an alternative scanner will be used. Throughout the study MRI methods will be adapted as appropriate to ensure optimal study results can be obtained.

FMD FMD will be offered to all participants in the main trial, but may be declined without affecting their participation in the main trial.

FMD on the brachial artery will be performed in the non-fistula arm on three visits (baseline, month 9 and month 12) using a Philips iE33 ultrasound machine (Phillips Medical Systems, United Kingdom) according to the guide-lines set by the International Brachial Artery Reactivity Task Force.[33] The brachial artery will be longitudinally imaged above the elbow using an 11.3-MHz probe. The image will be recorded for 2 minutes, followed by induction of forearm ischaemia by inflating a cuff below the elbow to 200 mmHg (or 50 mmHg above SBP, whichever is higher) for 5 minutes and deflating rapidly. The resulting reactive hyperaemia will be recorded for a further 2 minutes. After a rest period, the procedure will be repeated, with 0.4mg of glyceryl trinitrate being administered sublingually to determine endothelium-independent dilation. FMD will be expressed as per cent change in diameter relative to the baseline diameter at rest. Analysis of all FMDs will be performed on Brachial Analyser software (Medical Imaging Applications, LLC) by a single trained investigator (the clinical research fellow) to avoid inter-observer variability. This investigator will be blind to allocated treatments. Our intra-observer coefficient of variation for FMD is usually 5.2%. Two factors should ensure reliable results despite there being two sites : each patient will always be studied on the same equipment and wherever possible the same individual (the research fellow) will do all the tests and interpret them (blindly) at both sites. For further reassurance, a selection of blinded ultrasound scans will be re-analysed to ensure good reproducibility at each site and between sites.

Applanation Tonometry PWA will be offered to all participants in the main trial, but may be declined without affecting their participation in the main trial.

Pulse wave analysis (PWA) and PWV will be determined in the non-fistula arm by recording the radial waveforms and radial-carotid waveforms, respectively, at three visits (baseline, month 9 and month 12) using the Sphygmocor system. The central AIx will be corrected to a heart rate of 75 beats/min. Wherever possible, a single trained investigator (the clinical research fellow) who is blind to the allocated treatment will perform the PWA and PWV at both sites. We will also use bio-impedance at the same time to measure total body water in MRIs done at Glasgow sites.[21] . This will complement the end diastolic volume data from the MRI at both sites. In our index study, EDV fell but we did not know if this was due to afterload reduction or to a global fall in body water.[21] Bio-impedance will help determine this.

Research Blood tests Research bloods will be taken at baseline, week 6 and months 6, 9 and 12. Research bloods will include BNP, inflammatory markers and other markers of interest. Additional markers may be tested on the samples at a later date. The total amount of research blood taken at each visit will be no more than 30ml. We shall also seek consent for future ethically approved genetic testing which can be declined without affecting participation in the study. If agreement is given for this, 10mls of blood will be taken at the end of the study and anonymously stored - any subsequent analysis of these samples will be subject to approval of a Research Ethics Committee prior to analysis.

Adverse events Adverse events will be sought by symptom enquiry at each visit and by monitoring of routine blood samples.

ELIGIBILITY:
Inclusion Criteria:

* aged 18 years or over
* end stage renal disease (CKD stage 5 eGFR <15ml/min /1.73m2)
* been on haemodialysis for at least 3 months.

Exclusion Criteria:

* Known heart failure
* Left Ventricular Ejection Fraction <45%,
* active gout
* severe hepatic disease
* or on azathioprine, 6 mercaptopurine, theophylline.
* malignancy or other life threatening diseases,
* pregnant or lactating women
* any contraindication to MRI (claustrophobia, metal implants).
* with a planned (relative) kidney transplant,
* Patients who have participated in any other clinical trial within the previous 30 days will be excluded.
* Patients who are unable to give informed consent will also be excluded from this trial.
* Any other considered by a study physician to be inappropriate for inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2013-09; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
The primary outcome is to measure if allopurinol, induces a change in Left ventricular Mass Index in patients with ESRD when compared to placebo. | following 1 year of therapy

SECONDARY OUTCOMES:
To decide on optimum dosing regime of allopurinol in End Stage Renal Disease from pilot study | 6 weeks
  The dose of allopurinol required to reduce urate levels by 41% will be determined.
To measure any difference in endothelial function with allopurinol compared with placebo, measured by Flow Mediated Dilatation and Pulse Wave Analysis | following 1 year of therapy
To assess if the incidence of adverse events differs on allopurinol compared to placebo in patients with end stage renal disease | during course of 1 year of therapy
To measure any change in LV end systolic volume, LV end diastolic volume or LV ejection factor with allopurinol in ESRD patients compared with placebo. | Following 1 year of therapy
To measure changes in inflammatory blood markers, in ESRD with allopurinol compared with placebo. | Following 1 year of therapy
To measure changes in BP control as measured by clinic BP and 24hr BP monitoring with allopurinol compared with placebo | Following 1 year of therapy

CONTACTS AND LOCATIONS:
Overall Officials: Allan D Struthers, BSc, MD, FRCP, FESC, FRSE, Study Director — Centre for Cadiovascular Medicine, University of Dundee
Locations (3):
- United Kingdom (3):
  - NHS Greater Glasgow and Clyde, Glasgow, La
  - NHS Tayside, Dundee, Tayside
  - NHS Ayrshire and Arran, Crosshouse

REFERENCES:
- [Background] Kao MP, Ang DS, Gandy SJ, Nadir MA, Houston JG, Lang CC, Struthers AD. Allopurinol benefits left ventricular mass and endothelial dysfunction in chronic kidney disease. J Am Soc Nephrol. 2011 Jul;22(7):1382-9. doi: 10.1681/ASN.2010111185. Epub 2011 Jun 30. PMID 21719783